CLINICAL TRIAL: NCT05700734
Title: A Single-dose Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-retroviral Activity of MK-8510 Monotherapy in Anti-retroviral-naïve HIV-1 Infected Participants
Brief Title: MK-8510 Monotherapy for the Treatment of Anti-retroviral naïve Human Immunodeficiency Virus Type 1 (HIV-1) Infected Participants (MK-8510-002)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8510-002; MK-8510-002 (Other: Merck); 2021-006180-21 (EudraCT Number)
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: HIV-1; Human Immunodeficiency Virus 1; Immunodeficiency Virus Type 1, Human; Human Immunodeficiency Virus Type 1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Panel A: MK-8510 at dose level 1 (Experimental): Single oral dose of MK-8510 administered at dose level 1 (≤1800 mg) following a 10-hour fast. Dose level 1 shall not exceed 1800 mg.
  Interventions: Drug: MK-8510
- Panel B: MK-8510 at dose level 2 (Experimental): Single oral dose of MK-8510 administered at dose level 2 (≤2200 mg) following a 10-hour fast. Dose level 2 shall not exceed 2200 mg.
  Interventions: Drug: MK-8510
- Panel C: MK-8510 at dose level 3 (Experimental): Single oral dose of MK-8510 administered at dose level 3 (≤2200 mg) following a 10-hour fast. Dose level 3 shall not exceed 2200 mg.
  Interventions: Drug: MK-8510
- Panel D: MK-8510 at dose level 4 (Experimental): Single oral dose of MK-8510 administered at dose level 4 (≤2200 mg) following a 10-hour fast. Dose level 4 shall not exceed 2200 mg.
  Interventions: Drug: MK-8510

INTERVENTIONS:
Drug: MK-8510 — Single dose of MK-8510 administered as a tablet at a dose up to 2200 mg.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and anti-retroviral activity of MK-8510 monotherapy in anti-retroviral-naïve HIV-1 infected participants.

ELIGIBILITY:
Inclusion Criteria:

* Has HIV-1 infection, and is in good health based on medical history, physical examination, vital signs (VS) measurements, and laboratory safety tests.
* Has documented HIV-1 positive, as determined by a positive enzyme-linked immunosorbent assay (ELISA) or real-time quantitative polymerase chain reaction (QT-PCR) with confirmation (eg, Western Blot).
* Is anti-retroviral therapy (ART)-naïve, which is defined as:

  1. Having never received any anti-retroviral agent; or
  2. ART-experienced but has not received any ART for HIV-1 infection within 60 days; or
  3. Has received pre-exposure prophylaxis (PrEP) treatment prior to diagnosis of HIV-infection but has not received any PrEP within 30 days.
* Is willing to receive no other ART prior to Day 11 post-dose of the study.
* Has a body mass index (BMI) ≤35 kg/m2.

Exclusion Criteria:

* Has acute (primary) HIV-1 infection.
* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has remote history of uncomplicated medical events (eg, uncomplicated kidney stones, as defined as spontaneous passage and no recurrence in the last 5 years, or childhood asthma).
* Is mentally or legally incapacitated or has significant emotional problems.
* Has history of cancer (malignancy).
* Has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e, systemic allergic reaction) to prescription or nonprescription drugs or food.
* Has positive hepatitis B surface antigen (HBsAg).
* Has a history of chronic hepatitis C unless there has been documented cure and/or participant with a positive serologic test for hepatitis C virus (HCV) has a negative HCV viral load (VL).
* Had a major surgery and/or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Has participated in another investigational study within 4 weeks.
* Has a clinically significant abnormality on the electrocardiogram (ECG) performed at the pre-study visit.
* Has been committed to an institution by way of official or judicial order.
* Is under the age of legal consent or not capable of giving consent.
* Does not agree to follow the smoking restrictions as defined by the clinical research unit (CRU).
* Consumes greater than 3 servings of alcoholic beverages (1 serving is approximately equivalent to: beer [354 mL/12 ounces], wine [118 mL/4 ounces], or distilled spirits [29.5 mL/1 ounce]) per day.
* Consumes excessive amounts, defined as greater than 6 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day.
* Is a regular user of any illicit drugs (not including cannabis) or has an history of drug (including alcohol) abuse within approximately 12 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-17 (Estimated); Primary Completion 2024-02-14 (Estimated); Study Completion 2024-02-14 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Plasma HIV-1 Ribonucleic Acid (RNA) | Baseline and 168 hours post-dose
  The plasma HIV-RNA will be measured based on a longitudinal data analysis model containing fixed effects for dose level, and dose level by time interaction, and a random effect of MK-8510 (prodrug). The change from baseline for each dose level at 168-hours post baseline will be estimated from this model.
Percentage of Participants Who Experience an Adverse Event (AE) | Up to 36 days
  An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Percentage of Participants Who Discontinued from Study Due to an Adverse Event (AE) | Up to 36 days
  The percentage of participants who discontinue study due to an AE will be presented.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve of MK-8558 From Time 0 to 168 Hours (AUC0-168 hr) | At protocol specific timepoints up to 168 hours post-dose
  The AUC0-168 of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 12, 24, 48, 72, 120, 168 hours post-dose.
Area Under the Concentration-Time Curve of MK-8558 From Time 0 to last (AUC0-last) | At protocol specific time points up to 504 hours post-dose
  AUC0-last of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose.
Concentration at 168 Hours Post-dose (C168) of MK-8558 | 168 hours post-dose
  C168hr of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated.
Maximum Concentration (Cmax) of MK-8558 | At protocol specific time points up to 504 hours post-dose
  Cmax of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose.
Time to Maximum Plasma Concentration (Tmax) of MK-8558 | At protocol specific time points up to 504 hours post-dose
  Tmax of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose.
Half Life (t1/2) of MK-8558 | At protocol specific time points up to 504 hours post-dose
  t1/2 of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose.
Apparent Plasma Clearance of Drug After Extravascular Administration (CL/F) of MK-8558 | At protocol specific time points up to 504 hours post-dose
  CL/F of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose.
Apparent Volume of Distribution in the Terminal State After Extravascular Administration (Vz/F) of MK-8558 | At protocol specific time points up to 504 hours post-dose
  Vz/F of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose.
Terminal t1/2 of MK-8558 | At protocol specific time points up to 504 hours post-dose
  Terminal t1/2 of MK-8558 (active drug) after administration of MK-8510 (prodrug) in plasma will be calculated pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 12, 24, 48, 72, 120, 168, 240, 336, 504 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php